CLINICAL TRIAL: NCT06242873
Title: Transcutaneous Spinal Cord Stimulation in Children With Incomplete Spinal Cord Injury: Safety, Feasibility, and Efficacy.
Brief Title: Transcutaneous Spinal Cord Stimulation in Children With Incomplete Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Principal Investigator, Rebecca Martin, OTR/L, OTD, Asst Professor, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00300695
Record Dates: First submitted 2024-01-18; First posted 2024-02-05 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Spinal Cord Injuries
Keywords: Transcutaneous Spinal Cord Stimulation (TSCS)
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcutaneous Spinal Cord Stimulation and Gait Training (Experimental): Transcutaneous Spinal Cord Stimulation (TSCS), TSCS will be applied using an oval electrode placed midline on the skin on the back and two rectangular electrodes placed on the skin over the lower abdomen. There will be a small electrical current through those electrodes for 30 minutes.
  Interventions: Other: Gait training with/without TSCS
- Transcutaneous Spinal Cord Stimulation within a single session (Sham Comparator): Electrodes will be placed as they are in the Transcutaneous Spinal Cord Stimulation condition. Stimulation will be applied at subject's maximum intensity for 30 seconds and then discontinued.
  Interventions: Other: Gait training with/without TSCS

INTERVENTIONS:
Other: Gait training with/without TSCS — To assess the safety and impact of paired stimulation and training on gait in children with iSCI, participants will participate in 24 total sessions. Two sessions will involve assessment only and 22 sessions will include two hours of therapy. Sessions will occur at least three times per week, but may be scheduled as many as five times per week. In each session, participants will receive 60 minutes of treadmill training followed by strengthening, segmental task practice, and gait-based interventions. Participants will receive stimulation based on their group assignment (TSCS or sham).

SUMMARY:
Aim 1: Determine the safety and feasibility of administration of TSCS to children in a clinical setting. Participants will be randomly assigned to experimental (TSCS) or control (sham stimulation) groups. Both groups will receive eight-weeks of individualized gait training. We will measure adverse events, including pain and skin irritation, to determine safety as the primary outcome. Hypothesis 1: Administration of TSCS to children in a clinical setting will be safe based on similar safety outcomes as sham TSCS. Hypothesis 2: TSCS is feasible based on compliance to session interventions and long-term adherence to the protocol. Additionally, we will collect data on effort during sessions of both participant and therapist. We anticipate that the participants will report less effort in the experimental condition, as compared to the control and therapists will report equal effort across conditions.

Aim 2: Determine the neurophysiologic impact of TSCS within a single session. We hypothesize that participants will demonstrate increased volitional muscle activity and strength with TSCS as compared to sham stimulation. This will be assessed by surface EMG and hand-held dynamometry of the dominant-side quadriceps muscle during maximum volitional contraction (MVC), across multiple time points. Changes in EMG activity will indicate change in central excitability in response to stimulation.

Aim 3: Exploratory measurement of TSCS and gait training on walking function. We hypothesize that concurrent TSCS and gait training will augment walking function in children with iSCI, as compared to gait training with sham stimulation. In addition to outcomes defined above, participants will be assessed with clinically relevant outcome measures, to include the Timed Up and Go, 10-Meter Walk Test, Walking Index for Spinal Cord Injury II, and 6-Minute Walk Test. Data collected as part of this aim will elucidate trends in responder qualities and timeline of changes to inform future studies.

ELIGIBILITY:
Inclusion Criteria:

* Age 3-16
* ≥ 6 months post injury
* Non-progressive SCI
* American Spinal Injury Association Impairment Scale (AIS) Classification C or D AIS C is an incomplete classification where more than half of the key muscles below the neurological level have a muscle grade of 3 or less AIS D is an incomplete classification where more than half of the key muscles below the neurological level have a muscle grade of more than 3
* Neurologic level above T10
* Tolerates upright position for >30 minutes
* Able to advance one lower extremity (LE) when in standing, bracing and assistive device allowed
* Medically stable (no hospitalizations in last 3 mos.)
* Able to comply with The International Standards for neurological and functional Classification of Spinal Cord Injury (ISNCSCI) exam

Exclusion Criteria:

* Progressive Spinal Cord Injury or Disease (SCI/D) (Multiple Sclerosis, Acute Disseminated Encephalomyelitis, etc.)
* Active wounds
* Range of motion limits impacting gait training
* Cardiac pacemaker/defibrillator
* Active cancer diagnosis
* Absent LE reflexes
* Pregnancy

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) | session 1, 6, 12, 18, and 24 (5-8 weeks total)
  Measures walking function, balance, and mobility.
10-Meter Walk Test (10MWT) | session 1, 6, 12, 18, and 24 (5-8 weeks total)
  Measures walking speed.
Walking Index for Spinal Cord Injury II (WISCI II) | session 1, 6, 12, 18, and 24 (5-8 weeks total)
  Measures walking quality, including need for assistive device and physical assistance.
6-Minute Walk Test (6MWT) | session 1, 6, 12, 18, and 24 (5-8 weeks total)
  Measures walking endurance

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Martin, OTR/L, OTD, CPAM, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No